CLINICAL TRIAL: NCT04853732
Title: Pain Registry for Epidemiological, Clinical, and Interventional Studies and Innovation
Brief Title: PRECISION Pain Research Registry
Acronym: PRECISION
Status: Recruiting | Type: Observational
Sponsor: University of North Texas Health Science Center (Other)
Responsible Party: Sponsor
Other Study IDs: #2015-169
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — Saliva, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Low Back Pain Cases
- Chronic Pain-Free Controls

SUMMARY:
The PRECISION Pain Research Registry enrolls participants with chronic low back pain (cases) and participants who are free of chronic pain (controls) to study the epidemiology and management of chronic pain. The vision of the registry is to conduct research to provide a future for all unbounded by pain.

DETAILED DESCRIPTION:
Case participants complete case report forms at quarterly encounters, whereas control participants complete a case report form only at an initial encounter.

A series of validated or recommended research instruments are used or adapted by the registry for deployment in its case report forms. These may include some or all of the following at a given encounter:

* National Institutes of Health Minimum Dataset for Research on Chronic Low Back Pain
* Roland-Morris Disability Questionnaire
* Patient-Reported Outcomes Measurement Information System (PROMIS-29)
* History of Medical Conditions Inventory
* Pain Sensitivity Questionnaire
* Pain Catastrophizing Scale
* Pain Self-Efficacy Questionnaire
* Non-Pharmacological Treatments Inventory
* Pharmacological Treatments Summary
* Drug Adverse Events Index
* Physician Profile
* Physician Communication Behavior Questionnaire
* Physician Consultation and Relational Empathy Measure
* Patient Satisfaction Questionnaire (PSQ-18)

These instruments include measures that may serve as the independent or dependent variables in various substudies conducted by the registry over time, including observational studies (e.g., case-control studies, cohort studies) and randomized controlled trials.

The registry also maintains a biobank of biological specimens that have been collected from enrolled participants, including saliva and blood that may be used for DNA sequencing or biomarker analysis.

ELIGIBILITY:
Inclusion Criteria:

* Must reside within the contiguous 48 United States or District of Columbia
* Must provide a valid, government-issued identification with photo and birthdate
* Must have Internet access or telephone service to communicate with registry staff
* Must have sufficient English language proficiency to complete case report forms independently or with assistance from registry staff
* Must have a primary care physician or other physician who regularly provides health care
* Must provide the name, dose, and frequency of use of all current medications
* Case participants must have chronic low back pain
* Control participants must be free of any chronic pain and may include healthy volunteers

Exclusion Criteria:

* Must not be pregnant
* Must not reside in an institutional facility

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients seeking ongoing health care from a physician within the contiguous 48 United States or District of Columbia.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Case-Control Status | Upon registry enrollment
  Chronic Low Back Pain Case or Chronic Pain-Free Control

CONTACTS AND LOCATIONS:
Overall Officials: John C Licciardone, DO, MS, MBA, Principal Investigator — University of North Texas Health Science Center
Locations (1):
- University of North Texas Health Science Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Licciardone JC, Gatchel RJ, Aryal S. Effects of Opioids and Nonsteroidal Anti-Inflammatory Drugs on Chronic Low Back Pain and Related Measures: Results from the PRECISION Pain Research Registry. Tex Med. 2018 Oct 1;114(10):e1. PMID 30281768
- [Result] Licciardone JC, Schmitt ME, Aryal S. Empathy in Medicine Osteopathic and Allopathic Physician Interpersonal Manner, Empathy, and Communication Style and Clinical Status of Their Patients: A Pain Registry-Based Study. J Am Osteopath Assoc. 2019 Aug 1;119(8):499-510. doi: 10.7556/jaoa.2019.092. PMID 31305871
- [Result] Licciardone JC, Gatchel RJ. Osteopathic Medical Care With and Without Osteopathic Manipulative Treatment in Patients With Chronic Low Back Pain: A Pain Registry-Based Study. J Am Osteopath Assoc. 2020 Feb 1;120(2):64-73. doi: 10.7556/jaoa.2020.016. PMID 31985765
- [Result] Licciardone JC. Assessment of Longitudinal Clinical Outcome Measures for Chronic Low Back Pain over 12 Months. J Gen Intern Med. 2020 Dec;35(12):3733-3735. doi: 10.1007/s11606-020-05723-3. Epub 2020 Feb 19. No abstract available. PMID 32076968
- [Result] Licciardone JC, Pandya V. Use of Complementary Health Approaches for Chronic Low-Back Pain: A Pain Research Registry-Based Study. J Altern Complement Med. 2020 May;26(5):369-375. doi: 10.1089/acm.2019.0448. Epub 2020 Mar 11. PMID 32167785
- [Result] Licciardone JC, Pandya V. Prevalence and Impact of Comorbid Widespread Pain in Adults with Chronic Low Back Pain: A Registry-Based Study. J Am Board Fam Med. 2020 Jul-Aug;33(4):541-548. doi: 10.3122/jabfm.2020.04.190456. PMID 32675265
- [Result] Licciardone JC, Pandya V. Feasibility Trial of an eHealth Intervention for Health-Related Quality of Life: Implications for Managing Patients with Chronic Pain during the COVID-19 Pandemic. Healthcare (Basel). 2020 Oct 1;8(4):381. doi: 10.3390/healthcare8040381. PMID 33019676
- [Result] Licciardone JC. Demographic Characteristics Associated With Utilization of Noninvasive Treatments for Chronic Low Back Pain and Related Clinical Outcomes During the COVID-19 Pandemic in the United States. J Am Board Fam Med. 2021 Feb;34(Suppl):S77-S84. doi: 10.3122/jabfm.2021.S1.200352. PMID 33622822
- [Result] Licciardone JC. Impact of COVID-19 on utilization of nonpharmacological and pharmacological treatments for chronic low back pain and clinical outcomes. J Osteopath Med. 2021 Mar 29;121(7):625-633. doi: 10.1515/jom-2020-0334. PMID 33770828
- [Result] Licciardone JC, Aryal S. Patient-centered care or osteopathic manipulative treatment as mediators of clinical outcomes in patients with chronic low back pain. J Osteopath Med. 2021 Aug 3;121(10):795-804. doi: 10.1515/jom-2021-0113. PMID 34348426
- [Result] Licciardone JC. Preventing progression from chronic to widespread pain and its impact on health-related quality of life: a historical cohort study of osteopathic medical care. J Osteopath Med. 2021 Sep 23;122(1):21-29. doi: 10.1515/jom-2021-0105. PMID 34852185
- [Result] Licciardone JC, Ganta S, Goehring L, Wallace K, Pu R. Analysis of the Patient-Physician Relationship, Race, and Pain Control and Physical Function Among Adults With Chronic Low Back Pain. JAMA Netw Open. 2022 Jun 1;5(6):e2216270. doi: 10.1001/jamanetworkopen.2022.16270. PMID 35679045
- [Result] Licciardone JC, Aryal S. Nonadherence to Clinical Practice Guidelines for Opioid Prescribing in Patients with Chronic Low Back Pain: A Pain Research Registry-Based Study. J Am Board Fam Med. 2022 Jul-Aug;35(4):724-732. doi: 10.3122/jabfm.2022.04.210432. PMID 35896452
- [Result] Schultz MJ, Licciardone JC. The effect of long-term opioid use on back-specific disability and health-related quality of life in patients with chronic low back pain. J Osteopath Med. 2022 Aug 11;122(9):469-479. doi: 10.1515/jom-2021-0172. eCollection 2022 Sep 1. PMID 35950241
- [Result] Licciardone JC, McDonald H, Yablon M, Ngo W, Cunanan Garza KA, Aryal S. Optimizing chronic pain management through patient engagement with quality of life measures: a randomized controlled trial. J Osteopath Med. 2022 Aug 2;122(11):571-580. doi: 10.1515/jom-2021-0296. eCollection 2022 Nov 1. PMID 35918787
- [Result] Licciardone JC, Pandya V. Pain and functional recovery from chronic low back pain over 12 months: implications for osteopathic medicine. J Osteopath Med. 2022 Aug 24;122(12):623-630. doi: 10.1515/jom-2021-0288. eCollection 2022 Dec 1. PMID 35998917
- [Result] Licciardone JC, Beal J, Fakes N, Herron B, Jacobs C, Vasudevan A. The role of pain hypersensitivity in development of chronic widespread pain: a retrospective cohort study. Journal of Pain Management. January 2023;16(1):45-53.
- [Result] Licciardone JC, Patel S, Kandukuri P, Beeton G, Nyalakonda R, Aryal S. Patient Satisfaction With Medical Care for Chronic Low Back Pain: A Pain Research Registry Study. Ann Fam Med. 2023 Mar-Apr;21(2):125-131. doi: 10.1370/afm.2949. PMID 36973050
- [Result] Licciardone JC, Moore S, Fix K, Blair LG, Ta K. Osteopathic manipulative treatment of patients with chronic low back pain in the United States: a retrospective cohort study. J Osteopath Med. 2023 Feb 3;123(5):259-267. doi: 10.1515/jom-2022-0212. eCollection 2023 May 1. PMID 36732038
- [Result] Licciardone JC, Kellerlee J, Joseph M, Mohammad MB, Kim KG, Jain J, Aryal S. The process and outcomes of chronic low back pain treatment provided by osteopathic and allopathic physicians: a retrospective cohort study. J Osteopath Med. 2023 May 25;123(8):385-394. doi: 10.1515/jom-2023-0046. eCollection 2023 Aug 1. PMID 37225662
- [Result] Licciardone JC, Miller CL, Nazzal AJ, Hernandez CT, Nguyen LH, Aryal S. Racial Disparities in Opioid Use and Lumbar Spine Surgery for Chronic Pain and in Pain and Function Over 3 Years: A Retrospective Cohort Study. J Pain. 2024 Mar;25(3):659-671. doi: 10.1016/j.jpain.2023.09.018. Epub 2023 Sep 28. PMID 37777036
- See also: Participant screening site (cases) — http://www.unthsc.edu/research/precision-pain-research-registry/